CLINICAL TRIAL: NCT04712565
Title: Hard and Soft Tissue Maintenance Around Implants With a Sloped Configuration Without GBR in Comparison to a Conventional Neck Design With GBR-procedure: A Prospective Randomized Clinical Trial
Brief Title: Hard and Soft Tissue Maintenance Around Implants With a Sloped Configuration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32-514 ex 19/20
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astra Tech Implant System Profile EV (Experimental): Implants with sloped marginal configuration without bone augmentation are used.
  Interventions: Device: Astra Tech Implant System Profile EV
- Astra Tech Implant System EV (Active Comparator): Implants with regular neck design and GBR procedure fixed with two membrane pins will be used.
  Interventions: Device: Astra Tech Implant System EV

INTERVENTIONS:
Device: Astra Tech Implant System Profile EV — dental implant with a sloped neck configuration
  Arms: Astra Tech Implant System Profile EV
Device: Astra Tech Implant System EV — dental implant with a conventional neck configuration
  Arms: Astra Tech Implant System EV

SUMMARY:
This study is a controlled, randomized clinical trial over about 16-months (active phase). 40 patients in need of replacement of a single tooth with a minimal crestal bone width of 4 - 5mm and suitable for simultaneous GBR (Guided Bone Regeneration) procedure as well as at least a neighboring tooth on its mesial aspect will be consecutively recruited at the Department of Dental Medicine and Oral Health Graz. Volunteers will be screened and eligible subjects will be randomized to two different groups. In group 1 implants with regular neck design (Astra Tech Implant EV C, Dentsply Implants Manufacturing GmbH, Hanau, Germany) and GBR procedure (BioOss® and BioGide®, Geistlich, Wolhusen, Schweiz) fixed with two membrane pins (Hipp Medical AG, Kolbingen, Germany) will be used; in group 2 implants with sloped marginal configuration (Astra Tech Implant Profile EV C, Dentsply Implants Manufacturing GmbH, Hanau, Germany) without bone augmentation are used. The dimension of the bony defect and amount of lingual-buccal bone height discrepancy (max. 5mm) respectively bone width will be evaluated using a 3-D volume tomography (Planmeca ProMax® 3D Max, Planmeca, Helsinki, Finland), which is needed for digital planning (Simplant Planning Software, Leuven, Belgium) of the implant position, length and diameter as well.

DETAILED DESCRIPTION:
Digital scans will be done at first, 5th, 6th, 8th, and 10th visit to get the possibility to determine and compare volume changing and stability at augmented or not augmented implant sites during follow up visits.

According to standard procedure, patients will receive an antibiotic regime (Augmentin 1g, 2x1, GlaxoSmithKline, Vienna, Austria; in case of penicillin-allergy: DalacinC 300mg, 3x1, Pfizer, Vienna, Austria) starting one day prior surgery till 3 days after surgery. Before implant surgery patients are advised to rinse with a local antiseptic chlorhexidine gluconate solution (Chlorhexamed forte 2mg/ml, GlaxoSmithKline, Vienna, Austria). Articain is used for local anesthesia (Ultracain D-S forte with epinephrine 1:100.000, Sanofi Aventis, Vienna, Austria). These drugs are not object of the investigation. After flap elevation the lingual-buccal height discrepancy and bone width is measured using a periodontal probe. The implant surgery is done following the standard surgical protocol of implant placement of the Department of Dental medicine and Oral Health Graz using a pilot drill guide. After implant insertion the marginal bone level will be measured using a periodontal probe. Implant shoulder attends as a reference.

After implant insertion (Astra Tech Implant EV C or Astra Tech Implant Profile EV C, Dentsply Implants Manufacturing GmbH, Hanau, Germany), GBR (Astra Tech Implant EV C) and a healing period of approximately 3 months for both groups, the implants will be uncovered following the standard protocol of the Department of Dental medicine and Oral Health Graz, and titanium gingiva formers will be placed (non-investigational devices). After implant recovery the marginal bone level will be measured again using a periodontal probe. Implant shoulder attends as a reference.

All patients will receive CE-certified gingiva formers, which are used in the Department of Dental Medicine and Oral Health Graz and which are approved in Austria. 1 week after reentry the sutures will be removed and the digital impression (PrimeScan) for the CAD/CAM (Computer Aided Design /Computer Aided Manufacturing) manufactured single implant crowns using customized individual abutments (Atlantis, Mölndal, Sweden) will be done.

Radiographic examinations (single-tooth x-ray) will be done at implant recovery (3 months after implant placement, visit 6), visit 10 and visit 11.

A complete periodontal status (PD=probing depth, BOP= Bleeding on probing, PI= Plaque index) should be evaluated at the first visit (before implant placement). These parameters (PD, BOP, PI) as well as Papilla Index should be performed 8, 12, and 15 months after implant placement at implant and reference tooth site. In addition, PD and Papilla Index will be performed 4 months after implant placement (at time of integration of the implant crown). At the first visit, complete periodontal status will be evaluated to prove if the participant fulfills the inclusion criteria. During the following visits only reference teeth (neighboring tooth or teeth to the implant) and the implant site will be determined.

The soft tissue maintenance will be detected using the Papilla Index by Jemt (Jemt T, 1997) which assesses the size of interproximal gingival papillae adjacent to single implant restorations. Using this, one can determine the papilla remodeling between a dental implant and each neighboring tooth.

Intraoral photographs will be taken at every study visit (except suture removal), evaluating the esthetic outcome.

Oral Health Impact Profile (OHIP-G 14) will be done at the first visit and 12 months after implant placement. The Oral Health Impact Profile as a self-rating patient-centered instrument designed to assess the oral health-related quality of life within the last month. Especially, the following dimensions are captured by the OHIP-G 14: functional Limitation (e.g., "pronouncing any words because of problems with your teeth, mouth, dentures, or jaw?") and physical Pain (e.g., "Have you had painful aching in your mouth"). 14 questions are raised, which are answered using a rating scale from 0 (never) to 4 (very often).

A questionnaire evaluating patient satisfaction will be performed one week after implant surgery and 12 months after implant placement.

Visual analog scale (VAS) for subjective measurement of pain will be performed immediately and 1 week after implant placement using a combined VAS and numeric rating scale (NRS) The scale ranges from 0 (smiling face), which means no pain, to 10 (sad face), which means most pain imaginable).

GCP Statement: This study will be conducted in compliance with the principles of the Declaration of Helsinki, the ICH-GCP guidelines and in accordance with the relevant provisions of Austrian Medical Devices Act (MPG), the European Directive on implantable medical devices (90/385/EEC), the Styrian Hospitals Act (KALG), the Federal Law on hospitals (KAKuG), the EN-ISO standards 14155-1 and -2, EN ISO 14971, 10993 and all other ENISO eligible relevant legislations.

ELIGIBILITY:
Inclusion Criteria:

* Written consent after clarification
* capability of giving an informed consent
* good health as defined by the subjects medical history (no contraindications as described in the exclusion criteria below)
* age 18 years of age and over
* Good periodontal status: BOP < 20%, PI < 30%, no PD > 4mm
* No heavy smokers (< 10 cigarettes/day)
* At least 1 missing tooth in the premolar and molar region (in selected cases in the frontal area) either in the maxilla or in the mandible requiring implant therapy for reconstruction.
* implant site must present a buccal bone defect not extending a lingual-buccal or buccal-palatinal height discrepancy of 5mm and a sufficient bone width for simultaneously GBR procedure
* implant site must present at least a neighbouring tooth on its mesial aspect

Exclusion Criteria:

* Insufficient bone volume for implant placement requiring a sinus floor elevation or extensive bone augmentation
* Heavy Smokers (>10 cigarettes/day)
* Medication with a contraindication for implant therapy
* Skeletal immaturity
* Any active malignancy or ongoing treatment for malignancy
* An active infection at the operative site
* Contraindications to the class of drugs which are used at regular surgical procedures, e.g. known hypersensitivity or allergy to class of drugs or the investigational product, except penicillin-allergy
* Pregnancy
* unable or unwilling to return for follow-up visits for a period of at least 16 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
marginal bone level | 15 months
  measured by single tooth X-ray

SECONDARY OUTCOMES:
implant survival rate (ISR) in percent | 15 months
  measured in percent
clinical parameter: Probing depth | 15 months
  using a periodontal probe; in mm
clinical parameter: Bleeding on probing | 15 months
  in percent
clinical parameter: Plaque index | 15 months
  in percent
clinical parameter: Papilla index | 15 months
  Papilla Index (Jemt T, 1997), the index ranges from 0 to 4, while 2 and 3 indicate physiological outcome
patient satisfaction | 15 months
  no difference in patient satisfaction measured with OHIP G14 questionnaire. The following dimensions are captured by the OHIP-G 14: functional Limitation (e.g., "pronouncing any words because of problems with your teeth, mouth, dentures, or jaw?") and physical Pain (e.g., "Have you had painful aching in your mouth"). 14 questions are raised, which are answered using a rating scale from 0 (never) to 4 (very often).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Universtiy Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No
results will be shared by publishing an article

REFERENCES:
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Hof M, Pommer B, Strbac GD, Suto D, Watzek G, Zechner W. Esthetic evaluation of single-tooth implants in the anterior maxilla following autologous bone augmentation. Clin Oral Implants Res. 2013 Aug;24 Suppl A100:88-93. doi: 10.1111/j.1600-0501.2011.02381.x. Epub 2011 Dec 8. PMID 22150807
- [Background] Jemt T. Regeneration of gingival papillae after single-implant treatment. Int J Periodontics Restorative Dent. 1997 Aug;17(4):326-33. PMID 9497723
- [Background] Lekholm U, Adell R, Lindhe J, Branemark PI, Eriksson B, Rockler B, Lindvall AM, Yoneyama T. Marginal tissue reactions at osseointegrated titanium fixtures. (II) A cross-sectional retrospective study. Int J Oral Maxillofac Surg. 1986 Feb;15(1):53-61. doi: 10.1016/s0300-9785(86)80011-4. PMID 3083006
- [Background] Lorenzoni M, Pertl C, Wegscheider W, Keil C, Penkner K, Polansky R, Bratschko RO. Retrospective analysis of Frialit-2 implants in the augmented sinus. Int J Periodontics Restorative Dent. 2000 Jun;20(3):255-67. PMID 11203567
- [Background] Pietrokovski J, Massler M. Alveolar ridge resorption following tooth extraction. J Prosthet Dent. 1967 Jan;17(1):21-7. doi: 10.1016/0022-3913(67)90046-7. No abstract available. PMID 5224784
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Zuiderveld EG, Meijer HJ, Vissink A, Raghoebar GM. Outcome of Treatment with Single Implants in Preserved Versus Nonpreserved Alveolar Ridges: A 1-year Cohort Study. Int J Oral Maxillofac Implants. 2019 Nov/Dec;34(6):1457-1465. doi: 10.11607/jomi.7367. PMID 31711086
- [Background] Zumstein T, Schutz S, Sahlin H, Sennerby L. Factors influencing marginal bone loss at a hydrophilic implant design placed with or without GBR procedures: A 5-year retrospective study. Clin Implant Dent Relat Res. 2019 Oct;21(5):817-826. doi: 10.1111/cid.12826. Epub 2019 Aug 21. PMID 31432605
- [Result] Karasan D, Guncu MB, Ersu B, Canay S. Biomechanical Behavior of Implants with a Sloped Marginal Configuration. Int J Prosthodont. 2018 Nov/Dec;31(6):587-590. doi: 10.11607/ijp.5882. PMID 30408141
- [Result] Noelken R, Donati M, Fiorellini J, Gellrich NC, Parker W, Wada K, Berglundh T. Soft and hard tissue alterations around implants placed in an alveolar ridge with a sloped configuration. Clin Oral Implants Res. 2014 Jan;25(1):3-9. doi: 10.1111/clr.12079. Epub 2012 Dec 5. PMID 23210667